CLINICAL TRIAL: NCT03112226
Title: Effects of Ovarian Hormone Suppression on Vascular and Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 17-0092
Record Dates: First submitted 2017-04-07; First posted 2017-04-13 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Cognitive Impairment; Estrogen Deficiency; Menopause; Endothelial Dysfunction; Vascular Stiffness
Keywords: cognitive impairment; menopause; estrogen; functional MRI; executive function; endothelial function; arterial stiffness
MeSH Terms: conditions — Cognitive Dysfunction | interventions — LHRH, N-acetyl-(4-chlorophenylalanyl)(1)-(4-chlorophenylalanyl)(2)-tryptophyl(3)-arginyl(6)-alanine(10)-; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Estradiol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GnRHant + E2 (Active Comparator): Single dose of GnRH antagonist degarelix acetate for depot injection (80mg) Transdermal estradiol add-back; Climara patch, 0.075mg/day, weekly for 12 weeks
  Interventions: Other: GnRHant + E2
- GnRHant + Placebo (Placebo Comparator): Single dose of GnRH antagonist degarelix acetate for depot injection (80mg) Transdermal placebo patch, weekly for 12 weeks
  Interventions: Other: GnRHant + Placebo

INTERVENTIONS:
Other: GnRHant + E2 — GnRH antagonist with estradiol add-back
  Other Names: Degarelix acetate, Firmagon + Estradiol, Climara transdermal system
  Arms: GnRHant + E2
Other: GnRHant + Placebo — GnRH antagonist with placebo add-back
  Other Names: Degarelix acetate, Firmagon
  Arms: GnRHant + Placebo

SUMMARY:
Complaints about memory and thinking are common in women as they go through menopause. The female hormone estrogen is important for both the health of both the brain and the blood vessels. In Alzheimer's disease there is damage to the blood vessels in the brain. This study will look at how the loss of the female hormone estrogen affects brain function and the health of blood vessels.

ELIGIBILITY:
Inclusion Criteria:

* Stages of Reproductive Aging Workshop (STRAW+10) peak or late reproductive stage (-4, -3b or -3a)
* Healthy based on medical history, physical examination and standard blood chemistries
* Normotensive (resting blood pressure <140/90 mmHg)
* Normoglycemia (fasting glucose <110mg/dl and hemoglobin A1c<6.5%)
* Non-smoker (for at least 12 months)

Exclusion Criteria:

* Serum Follical Stimulating Hormone (FSH) >25mIU/mL measured during the first 5 days of the menstrual cycle
* Use of hormonal therapy within the past 3 months
* Use of antihypertensive or lipid-lowering medications
* Pregnant or lactating, or planning to become pregnant during the study period
* Known hypersensitivity to any of the study medications
* Abnormal vaginal bleeding
* History of venous thromboembolism or hormone-sensitive cancer
* History of neurologic disease or major psychiatric illness
* History of diagnosed learning disability or less than high-school education
* Contraindication to Magnetic Resonance Imaging (MRI) scanning
* Depression (Center for Epidemiological Studies - Depression (CESD) score >16)
* Significant cognitive impairment (Mini Mental State Examination (MMSE) score <27)
* Severe osteopenia or osteoporosis (proximal femur or lumbar spine T-score < -2.0)
* Body Mass Index (BMI) >40kg/m2

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2020-06-06 (Actual); Study Completion 2020-06-21 (Actual)

PRIMARY OUTCOMES:
Changes in Prefrontal cortex brain activation | Baseline, 3 months
  Changes in patterns of brain activation in the prefrontal cortex using functional magnetic resonance imaging (fMRI) during a task of working memory will be measured at baseline and 3 months

SECONDARY OUTCOMES:
Changes in Endothelial function | Baseline, 3 months
  Endothelial function will be measured using brachial artery flow-mediated dilation at baseline and 3 months
Changes in Arterial stiffness | Baseline, 3 months
  Carotid artery compliance will be measured using ultrasound at baseline and 3 months
Changes in Executive cognitive function | Baseline, 3 months
  Changes in executive cognitive function on a battery of neuropsychological tests will be measured at baseline and 3 months

OTHER OUTCOMES:
Changes in Mitochondrial dysfunction | Baseline and 3 months
  Measures of mitochondrial function including dynamics (fusion, fission), antioxidant defense and biogenesis will be measured in mitochondria isolated from peripheral blood mononuclear cells at baseline and 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Kerry L Hildreth, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Colorado Boulder Intermountain Neuroimaging Consortium, Boulder, Colorado

IPD SHARING:
Plan to Share IPD: No